CLINICAL TRIAL: NCT02048280
Title: Comparing NAVA Levels in Intubated and Recently Extubated Neonates to Determine Optimal Non-invasive Ventilatory Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TCH02
Record Dates: First submitted 2014-01-13; First posted 2014-01-29 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Other Specified Respiratory Problems in Fetus or Neonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intubated (Experimental): NAVA level from 0.1 to 3
  Interventions: Procedure: NAVA level; Other: NAVA level

INTERVENTIONS:
Procedure: NAVA level — Peak inspiratory pressure will be measured at each NAVA level
Other: NAVA level — Increase NAVA level every 3 minutes

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is a mode of mechanical ventilation that uses the diaphragm's normal electrical activity to deliver a mechanically supported breath. The amount of support provided is determined in part by the NAVA level, where a higher NAVA level will provide higher level of support and unload more of the work of the diaphragm. The purpose of this study is to compare the optimal NAVA level in neonates while on mechanical ventilation while intubated and after being extubated.

DETAILED DESCRIPTION:
Baseline measurements will be taken. The NAVA titration study will then be done. The NAVA level will be set at a starting value of 0.1 cm H2O/mcV and systematically increased by 0.5 cm H2O/mcV every three minutes to a maximum of 3 cmH2O/mcV. Once the NAVA titration study has been completed, the patient will be extubated. There will be a stabilization period following extubation (15-30 minutes), and then the NAVA titration study will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Neonates on NAVA ventilation

Exclusion Criteria:

-

Ages: 23 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in breakpoint in intubated and extubated patients | 20 minute study pre and post extubation
  NAVA titration study will be done pre and post extubation to determine and then compare the breakpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Stein, MD, Principal Investigator — Promedica Toledo Childrne's Hospital
Locations (1):
- Promedica Toledo CHildren's Hospital NICU, Toledo, Ohio, United States